CLINICAL TRIAL: NCT06553157
Title: Evaluation of the Effect of Statins on the Incidence of Side Effects of Platinum Based Chemotherapy in Patients With Solid Tumors
Brief Title: Statins Effect on Incidence of Side Effects of Platinum Based Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Collaborators: Minia University Hospital (Other)
Responsible Party: Principal Investigator, Noha Hassan Mohamed Helmy, Teaching asistant in clinical pharmacy department, Faculty of Pharmacy, Minia university, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Statins in ototoxicity
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumors; Ototoxicity
Keywords: platinum based chemotherapy; Cisplatin; adverse effects; ototoxicity; statins
MeSH Terms: conditions — Ototoxicity | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): no intervention
- intervention group (Experimental): study drug once daily for treatment period
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Statin — Statins are drugs known to help lower total cholesterol and reduce the risk of a heart attack or stroke. Statins include atorvastatin , fluvastatin , lovastatin , pitavastatin , pravastatin, rosuvastatin and simvastatin.
  Other Names: atorvastatin
  Arms: intervention group

SUMMARY:
Platinum based chemotherapy (mainly Cisplatin) is known to cause a variety of adverse effects, including Ototoxicity and nephrotoxicity. Ototoxicity is estimated to affect about 36% of adult patients treated with cisplatin, many therapeutic interventions have been studied to reduce the risk of developing ototoxicity from Cisplatin treatment, Statins have been studied in animals and have shown promising results, this study is aimed to explore the effect of statins on the incidence of ototoxicity in humans.

DETAILED DESCRIPTION:
Cisplatin and other platinum salt agents, including carboplatin and oxaliplatin, are widely used chemotherapy agents in patients with solid malignancies. These agents remain the backbone of treatment for ovarian, cervical, testicular, non-small-cell lung, bladder, and head and neck cancers. It is estimated that more than 500,000 patients diagnosed with these cancers annually in the United States could be candidates for treatment with cisplatin. However, adverse effects such as ototoxicity, neurotoxicity, and nephrotoxicity can sometimes limit their use. The incidence of ototoxicity induced by cisplatin has been estimated to be 36% of adult patients with cancer and 40%-60% of pediatric patients. Ototoxicity can be vestibular or cochlear toxicity or both, which can manifest as tinnitus (ringing in the ear), ear pain, and frank hearing loss.

The receipt of cisplatin is associated with a 5-fold increase in the risk of hearing impairment, and the incidence and severity are cumulative with exposure. Ototoxicity can manifest as tinnitus, hearing loss in the high-frequency range (4,000 to 8,000 Hz), or at late stages, a decreased ability to hear in the lower-frequency normal conversation range. It can occur during or after treatment and can be unilateral or bilateral affect both ears. Usually, hearing loss can start at higher frequencies in the beginning and can be permanent. In fact, severe ototoxicity with deafness has been reported even after a single cycle of cisplatin. Hence, monitoring and early identification of cisplatin-induced hearing loss are crucial to prevent detrimental impact on hearing and thereby the quality of life (QoL). Children affected by hearing loss have a poorer QoL as evident from their ability to communicate and interact with family and peers, their independence, and emotional well-being.The negative impact of hearing impairment on the patients' health-related QoL including social isolation, anxiety, and depression is well supported by a large body of evidence.

In the literature, two studies were found exploring the effect of statins on the incidence of ototoxicity induced by cisplatin, one retrospective study found that patients who used statins concurrently with their cisplatin chemotherapy had a lower incidence of developing ototoxicity, similar results were proven by a study conducted on mice that found that lovastatin protects against development of ototoxicity resulting from cisplatin therapy , a randomized controlled trial exploring the effect of statins on ototoxicity is needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients will receive platinum based chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients receiving vitamin/ supplementation drugs that interfere with the study intervention.
* Patients with contraindications to statins including acute liver failure or decompensated cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
change in hearing as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) using Audiometry as a tool | 3 months after end of treatment
  grade 1:Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6, and 8 kHz audiogram): Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear.
  grade 2: enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6, and 8 kHz audiogram): Threshold shift of >25 dB averaged at 2 contiguous test frequencies in at least one ear.
  grade 3: enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6, and 8 kHz audiogram): Threshold shift of >25 dB averaged at 3 contiguous test frequencies in at least one ear; therapeutic intervention indicated.
  grade 4: Decrease in hearing to profound bilateral loss (absolute threshold >80 dB HL at 2 kHz and above); nonservicable hearing
adapted version of the Speech, Spatial and Qualities of Hearing Scale 12 (SSQ12) | 3 months after end of treatment
  adapted version of the Speech, Spatial and Qualities of Hearing Scale 12 (SSQ12)

CONTACTS AND LOCATIONS:
Overall Officials: Noha H. Helmy, Masters, Principal Investigator — Department of Clinical Pharmacy, Faculty of Pharmacy, Minia University; Fatma M. Mady, Professor, Study Chair — Pharmaceutics Department, Faculty of Phramacy, Minia university; Nada H. Ali Sholkami, PhD, Study Director — Department of Clinical Oncology, Faculty of Medicine, Minia University; Eman M. Sadek, PhD, Study Director — Deaprtment of Clinical Pharmacy, Faculty of Pharmacy, Minia university; Dalia F. Mohammed Fahim, PhD, Study Director — Department of ENT, Audio-Vestibular Unit, Faculty of Medicine,Minia University
Locations (1):
- Minia University hospital, department of oncology and nuclear medicine, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez K, Spielbauer KK, Rusheen A, Wang L, Baker TG, Eyles S, Cunningham LL. Lovastatin protects against cisplatin-induced hearing loss in mice. Hear Res. 2020 Apr;389:107905. doi: 10.1016/j.heares.2020.107905. Epub 2020 Feb 6. PMID 32062294
- [Background] Fernandez KA, Allen P, Campbell M, Page B, Townes T, Li CM, Cheng H, Garrett J, Mulquin M, Clements A, Mulford D, Ortiz C, Brewer C, Dubno JR, Newlands S, Schmitt NC, Cunningham LL. Atorvastatin is associated with reduced cisplatin-induced hearing loss. J Clin Invest. 2021 Jan 4;131(1):e142616. doi: 10.1172/JCI142616. PMID 33393488
- [Background] Dalton DS, Cruickshanks KJ, Klein BE, Klein R, Wiley TL, Nondahl DM. The impact of hearing loss on quality of life in older adults. Gerontologist. 2003 Oct;43(5):661-8. doi: 10.1093/geront/43.5.661. PMID 14570962